CLINICAL TRIAL: NCT03717935
Title: Oral Amino Acid Nutrition to Improve Glucose Excursions in PCOS
Acronym: ORANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-0803
Record Dates: First submitted 2018-06-15; First posted 2018-10-24 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Polycystic Ovarian Syndrome; Obesity; Hepatic Steatosis
Keywords: hepatic de novo lipogenesis
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Fatty Liver | interventions — Amino Acids, Essential; Excitatory Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational drug pharmacy will performed randomization and dispense the EAA or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Essential Amino Acid (EAA) Supplement (Experimental): 4 weeks: Essential Amino Acid Supplement- 15g 2/day
  Interventions: Dietary Supplement: Essential Amino Acid (EAA) Supplement; Other: Placebo
- Placebo (Placebo Comparator): 4 weeks: Placebo- 15g 2/day
  Interventions: Dietary Supplement: Essential Amino Acid (EAA) Supplement; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Essential Amino Acid (EAA) Supplement — Powder supplement
Other: Placebo — Powder that will be similar to the essential amino acid supplement

SUMMARY:
The Investigators will measure hepatic glucose and fat metabolism in obese girls with Polycystic Ovarian Syndrome (PCOS) and hepatic steatosis (HS) after taking 4 weeks of an essential amino acid (EAA) supplement or placebo and test whether the EAA supplement can improve hepatic glucose metabolism in these girls.

DETAILED DESCRIPTION:
Girls with Polycystic Ovarian Syndrome (PCOS) and hepatic steatosis (HS) will complete a 12 week double-blinded placebo controlled cross-over study with 4 weeks each of an essential amino acid (EAA) supplement and placebo, and will complete metabolic studies after each intervention. There will be a 4 week wash out period in-between. The metabolic tests after each intervention (EAA/placebo) will include an oral sugar tolerance test (OSTT) and an oral U-C13 glycerol tracer that is paired with Nuclear Magnetic Resonance (NMR) isotopomer analysis of serum samples to describe flux through the hepatic pentose phosphate pathway, tricarboxylic acid (TCA) cycle and fatty acid synthesis pathways in girls with PCOS and HS. Hepatic steatosis will be measured with magnetic resonance Imaging (MRI) and hepatic phosphate concentrations with magnetic resonance (MR) spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Females
2. Ages 12-21
3. Sedentary- less than 2 hours of moderate (jogging, swimming etc) exercise a week.
4. BMI equal or greater than the 90th percentile for age and gender
5. PCOS per the most stringent NIH criteria adapted for adolescents (irregular menses >24 months post-menarche and clinical or biochemical hypertestosteronemia)
6. HS per FibroScan ultrasound, with CAP score of >225 (will be measured at screening visit)

Exclusion Criteria:

1. Use of medications known to affect insulin sensitivity: metformin, oral glucocorticoids within 10 days, atypical antipsychotics, immunosuppressant agents, HIV medications, hormonal contraception. Dermal patch or vaginal ring contraception methods.
2. Currently pregnant or breastfeeding women. Development of pregnancy during the study period will necessitate withdrawal from the study.
3. Severe illness requiring hospitalization within 60 days
4. Diabetes, defined as Hemoglobin A1C > 6.4%
5. BMI percentile less than the 90th percentile for age and sex. Weight >325 lbs or <84 lbs.
6. Anemia, defined as Hemoglobin < 11 mg/dL
7. Diagnosed major psychiatric or developmental disorder limiting informed consent
8. Implanted metal devices that are not compatible with MRI
9. Use of blood pressure medications
10. Known liver disease other than NAFLD or AST or ALT >125 IU/L

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Cree-Green, MD, PhD, Principal Investigator — Department of Endocrinology
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be shared with IRB approved personnel.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a crossover study. There were a total of 27 participants enrolled in the study. Four participants were never randomized: 3 screen failed and 1 of withdrew. Two participants withdrew after completing the placebo phase of the study
Groups:
- Essential Amino Acid (EAA) Supplement Followed by Placebo: Participants completed: 4 weeks of Essential Amino Acid Supplement- 15g 2/day followed by 4 weeks washout period and then 4 weeks of Placebo- 15g 2/day.
- Placebo Followed by Essential Amino Acid (EAA) Supplement: Participants completed: 4 weeks of Placebo- 15g 2/day followed by 4 weeks washout period and then 4 weeks of Essential Amino Acid Supplement- 15g 2/day.
Period: Overall Study
Arm/Group | Essential Amino Acid (EAA) Supplement Followed by Placebo | Placebo Followed by Essential Amino Acid (EAA) Supplement
Started | 11 | 12
Completed | 11 | 10
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Essential Amino Acid (EAA) Supplement vs Placebo: All study participants completed two 4-week phases of the study in random order with a washout period in between each phase of the study. Each phase consisted of either: 4 weeks of Essential Amino Acid Supplement- 15g 2/day followed by 4 weeks: Placebo- 15g 2/day or vice versa. We are comparing the differences in the essential amino acid vs placebo between all participants.
Arm/Group | All Study Participants: Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.67 (1.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Fat Fraction
Description: Hepatic Fat Fraction measured after completing placebo and amino acid therapy measured with MRI, and calculated via the Dixon method as the proton density hepatic fat fraction, which ranges from 0-75%. Greater than 5% is considered extra fat
Time Frame: 4 weeks after completing the first intervention, and approximately 8 weeks later (4 weeks washout and 4 weeks of second intervention)
Population: adolescent girls with PCOS
Measure: Median (Inter-Quartile Range); unit: percent hepatic fat
Groups:
- Essential Amino Acid (EAA) Supplement vs Placebo: Participants completed two 4-week phases of the study in random order with a washout period in between each phase of the study. Each phase consisted of either: 4 weeks of Essential Amino Acid Supplement- 15g 2/day followed by 4 weeks: Placebo- 15g 2/day or vice versa. We are comparing the differences in the essential amino acid vs placebo.
  Results reported are measured after completing each phase of the study placebo vs EAA
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 21
percent hepatic fat
  After 4 weeks of Placebo | 8 [4.1 to 15.9]
  After 4 weeks of EAA | 7.3 [3.9 to 16]

2. Secondary Outcome: Rate of De Novo Lipogenesis
Description: The rate of overnight de novo lipogenesis will be measured utilizing stable isotope methods with deuterated water, and expressed as the rate of newly synthesized lipids in the serum triglyceride fraction measured after 4 weeks of placebo and after 4 weeks of EAA intervention.
Time Frame: 4 weeks after the first intervention, and approximately 8 weeks later (4 weeks washout and 4 weeks of second intervention)
Population: We were only able to obtain results for this outcome for 19 participants in the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 19
mg/dL
  After 4 weeks of Placebo | 9.60 (6.10)
  After 4 weeks of EAAs | 6.55 (5.52)

3. Secondary Outcome: Evaluation of Mitochondrial Function
Description: Mitochondrial function will be assessed via change in direct hepatic carbon flux in newly synthesized triglycerides (TGs) using an oral sugar tolerance test with an oral UC13 glycerol tracer after each intervention. Data from 180 minutes post-tracer drink is shown below. A higher direct percent means less indirect futile cycling through the TCA cycle.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent direct TG synthesis
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 19
percent direct TG synthesis
  After 4 weeks of Placebo | 82.4 (2.5)
  After 4 weeks of EAAs | 82.5 (2.8)

4. Secondary Outcome: Hepatic Phosphate Profile After EAA and Placebo Supplement
Description: hepatic phosphate profile via 31 Phosphorus MR spectroscopy after each intervention
  Hepatic phosphate relative concentrations will be measured with 31 phosphorus magnetic resonance spectroscopy after each intervention. The Total phosphate (TP) concentration will be reported after each intervention and the ratio of the following phosphate metabolites will be reported over the total phosphate concentration: Phosphodiesterase (PDE), phosphomonoester (PME), Adenosine triphosphate (ATP), Inorganic Phosphate (Pi),Nicotinamide adenine dinucleotide phosphate (NADPH), Uridine diphosphate glucose (UDPG)
Time Frame: as for outcome 2
Population: We were only able to analyze 18 participants p-31 spectroscopy due to the quality of the spectra.
Measure: Mean (Standard Deviation); unit: Ratio over Total Phosphate Concentration
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 18
Ratio over Total Phosphate Concentration
  PDE/TP after EAA | 0.19670949 (0.049409797)
  PDE/TP after Placebo | 0.186460069 (0.034108394)
  PME/TP after EAA | 0.073640887 (0.036231645)
  PME/TP after Placebo | 0.074795509 (0.023577971)
  ATP/TP after EAA | 0.561426026 (0.088487664)
  ATP/TP after Placebo | 0.564456782 (0.053141701)
  Pi/TP after EAA | 0.056107611 (0.022628913)
  Pi/TP after Placebo | 0.064446077 (0.034944194)
  NADPH/TP after EAA | 0.085554177 (0.033832954)
  NADPH/TP after Placebo | 0.069352473 (0.035960915)
  UDPG/TP after EAA | 0.02656181 (0.017694541)
  UDPG/TP after Placebo | 0.040489089 (0.01814369)

5. Secondary Outcome: Whole Body Insulin Sensitivity
Description: Participants will undergo a 75 gram oral glucose tolerance test, and whole body insulin sensitivity will be expressed as Si, calculated via the oral minimal model using 4 hour glucose and insulin data during the OGTT after each phase of the study (placebo vs EAA).
Time Frame: as for outcome 2
Population: Only 20 participants analyzed because the OMM model cannot be run if we have missing insulin or glucose values during the oral sugar tolerance test.
Measure: Mean (Inter-Quartile Range); unit: dl/kg/min per microU/ml
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 20
dl/kg/min per microU/ml
  After 4 weeks of Placebo | 0.00026 [0.0002 to 0.00046]
  After 4 weeks of EAA | 0.00025 [0.00021 to 0.00043]

6. Secondary Outcome: Change in Adipose Insulin Sensitivity
Description: Change from baseline of adipose insulin sensitivity will be calculated as the percent suppression of free fatty acids (FFAs) during the oral glucose tolerance test.
Time Frame: as for outcome 2
Population: This measure was completed by 22 participants in the placebo phase of the study and 20 in the EAA phase of the study
Measure: Mean (Standard Deviation); unit: percent suppression FFAs
Groups:
- Essential Amino Acid (EAA) Supplement vs Placebo: Participants completed two 4-week phases of the study in random order with a washout period in between each phase of the study. Each phase consisted of either: 4 weeks of Essential Amino Acid Supplement- 15g 2/day followed by 4 weeks: Placebo- 15g 2/day or vice versa. We are comparing the differences in the essential amino acid vs placebo.
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 22
percent suppression FFAs
  4 weeks of Placebo | 91.15 (3.48)
  4 weeks of EAAs: number analyzed (Participants) | 20
  4 weeks of EAAs | 91.11 (4.18)

7. Secondary Outcome: Sleep Duration
Description: Sleep duration will be assessed completing placebo and essential amino acid therapy using home actigraphy. Change in sleep duration reported in minutes.
Time Frame: as for outcome 2
Population: Out of these 3 participants 2 did not complete their EAA phase for this measurement, so results reported for EAA only include 21 participants.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 21
minutes
  After 4 weeks of placebo | 390 (64)
  After 4 weeks of EAA | 340.7 (95.5)

8. Secondary Outcome: Apnea Hypopnea Index (AHI)
Description: Apnea Hypopnea Index (AHI) will be measured using WatchPAT after each intervention. In children and adolescents the scale that will be used is AHI>5 is considered mild sleep apnea. The higher the AHI, indicates more severe sleep apnea.
  The AHI is the number of times you have apnea or hypopnea during one night, divided by the hours of sleep.
  Normal sleep: An AHI of fewer than five events, on average, per hour Mild sleep apnea: An AHI of five to 14 events per hour Moderate sleep apnea: An AHI of 15 to 29 events per hour Severe sleep apnea: An AHI of 30 or more events per hour
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 21
events per hour
  After 4 weeks of Placebo | 14.99 (7.00)
  After 4 weeks of EAA | 17.04 (8.44)

9. Secondary Outcome: Amino Acid Metabolomics: Alanine, Glutamate, Leucine, Valine Levels After 4 Weeks of Placebo and 4 Weeks of EAAs
Description: Targeted amino acid metabolomics will be performed after each intervention and the levels of these 4 amino acids will be reported after each intervention.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: micro molar
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 21
micro molar
  Alanine after Placebo | 420 (120)
  Glutamate after Placebo | 49 (20)
  Leucine after Placebo | 91 (16)
  Valine after Placebo | 303 (36)
  Alanine after EAAs | 385 (116)
  Glutamate after EAAs | 54 (21)
  Leucine after EAAs | 88 (20)
  Valine after EAAs | 284 (46)

10. Secondary Outcome: Lipid Metabolomics: 16n1
Description: Targeted lipid metabolomics will be performed after each intervention to measure 16n1 lipids after completing 4 weeks of essential amino acid therapy and 4 weeks of placebo.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: micro molar
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 21
micro molar
  After 4 weeks of Placebo | 87 (45)
  After 4 weeks of EAAs | 88 (32)

11. Secondary Outcome: Bile Acid Metabolomics: Sphingosine-1-phospate After 4 Weeks of Placebo and 4 Weeks of EAAs
Description: Targeted bile acid metabolomics will be performed after each intervention to measure levels of sphingosine-1-phospate
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: micro molar
Arm/Group | Essential Amino Acid (EAA) Supplement vs Placebo
Number analyzed (Participants) | 21
micro molar
  After 4 weeks Placebo | 1334 (194)
  After 4 weeks EAAs | 1294 (281)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- All Participants: Essential Amino Acid (EAA) Supplement vs Placebo: All participants completed two 4-week phases of the study in random order with a washout period in between each phase of the study. Each phase consisted of either: 4 weeks of Essential Amino Acid Supplement- 15g 2/day followed by 4 weeks: Placebo- 15g 2/day or vice versa. We are comparing the differences in the essential amino acid vs placebo.
Arm/Group | All Participants: Essential Amino Acid (EAA) Supplement vs Placebo
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT03717935/Prot_SAP_000.pdf